CLINICAL TRIAL: NCT04755075
Title: A Phase 1 Study To Assess The Effect Of Hepatic Impairment On The Pharmacokinetics Of Surufatinib
Brief Title: Surufatinib Hepatic Impairment Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-012-00US2
Record Dates: First submitted 2021-02-04; First posted 2021-02-15 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Subjects with Normal Hepatic Function: All patients to receive study drug (Surufatinib 250mg) on Day 1
  Interventions: Drug: Surufatinib
- Cohort 2 (Experimental): Subjects with Moderate Hepatic Impairment: All patients to receive study drug (Surufatnib 250mg) on Day 1
  Interventions: Drug: Surufatinib
- Cohort 3 (if enrolled) (Experimental): Subjects with Mild Hepatic Impairment: All patients to receive study drug (Surufatnib 250mg) on Day 1
  Interventions: Drug: Surufatinib

INTERVENTIONS:
Drug: Surufatinib — Subjects to receive Surufatinib 250 mg on Day 1
  Other Names: HMPL-012
  Arms: Cohort 1
Drug: Surufatinib — Subjects to receive Surufatinib 250 mg on Day 1
  Other Names: HMPL-012
  Arms: Cohort 2; Cohort 3 (if enrolled)

SUMMARY:
An open-label, multicenter, single-dose, single-period, sequential study to determine the effect of hepatic impairment on the PK of surufatinib.

DETAILED DESCRIPTION:
This is a phase 1, open-label, multicenter, single-dose, single-period, sequential study with the primary objective of determining the effect of moderate and mild hepatic impairment on the PK of surufatinib. The secondary objective is to evaluate the safety in subjects with moderate and mild (if enrolled) hepatic impairment and subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Male or female between 18 and 75 (inclusive)
* Subject has BMI >18 and ≤40 kg/m^2 and body weight not ≤50 kg at screening.
* The subject is a non-smoker or light smoker who smokes no more than 10 cigarettes, 2 cigars, 2 pipes, or other nicotine equivalents (eg, vape, snuff, gum) of tobacco per day; willing to limit smoking during the treatment period to 4 cigarettes or 1 cigar per day.
* Females of non-childbearing potential or surgically sterile
* Males who have not had a successful vasectomy and are partners of women of childbearing potential must use, or their partners must use, a medically acceptable method of contraception starting for at least 1 menstrual cycle prior to and throughout the entire study period, and for 2 weeks after the last dose of study drug. Those with partners using hormonal contraceptives must also use an additional approved method of contraception such as a condom with spermicide. Males who have had a successful vasectomy (confirmed azoospermia, documentation needed) require no additional contraception. No sperm donation is allowed during the study period and for 90 days after study drug discontinuation.

Subjects with Hepatic Impairment

* For moderate hepatic impairment, the subject must have a Child-Pugh score of 7 to 9. For mild hepatic impairment, the subject must have a Child-Pugh score of 5 to 6.
* The subject must have no clinically significant change in disease status within the last 30 days before screening.
* If diabetic, the subject must have the disease controlled
* Subjects with ascites must not have a paracentesis within 3 months of screening.
* The subject must have blood pressure between 90 and 160 mm Hg systolic, inclusive, and not higher than 100 mm Hg diastolic.

Subjects with Normal Hepatic Function

* The subject must be without hepatic disease and have normal hepatic function
* The subject must be in good health
* The subject must have blood pressure between 95 and 150 mm Hg systolic, inclusive, and no higher than 90 mm Hg diastolic

Exclusion Criteria:

All Subjects

* The subject has evidence of clinically significant cardiovascular, GI, renal, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities.
* The subject has a known history of any GI surgery or any condition possibly affecting drug absorption.
* The subject has a clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to the first dose.
* The subject has a clinically significant ECG abnormality
* The subject has been diagnosed with acquired immune deficiency syndrome (AIDS), or tests positive for human immunodeficiency virus (HIV).
* The subject has participated in a clinical study of another drug before dosing, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks before Day 1, whichever is longer, or is currently enrolled in another clinical study.
* The subject has consumed grapefruit, starfruit, Seville oranges, or their products within 7 days prior to the first dose.
* The subject has consumed herbal preparations/medications, including, but not limited to, kava, ephedra (ma huang), Ginkgo biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng, within 7 days prior to the first dose.
* The subject has received blood or blood products within 8 weeks, or donated blood or blood products within 8 weeks prior to the first dose, or donated double red cells within 16 weeks prior to the first dose.
* The subject has used any drug that is a strong inhibitor or inducer (including St. John's wort) of CYP3A or P-gp within 2 weeks prior to first dose or will require use during study treatment period.
* The subject is allergic to the study drug or to any of its excipients.
* Female subjects who are pregnant or planning to become pregnant, lactating, or breastfeeding.
* The subject has used a proton pump inhibitor (PPI) within 4 days prior to the first dose or a histamine 2 (H2) receptor antagonist (H2 blocker) within 2 days prior to the first dose.

Subjects with Hepatic Impairment

* The subject has clinically significant vital sign abnormalities at screening or baseline.
* The subject has used acetaminophen at doses >1 g/day within 2 weeks prior to study drug administration.
* The subject has a history or current diagnosis of uncontrolled or significant cardiac disease indicating significant risk of safety for participation in the study
* The subject has Gilbert's syndrome, liver transplant, Wilson's disease, autoimmune liver disease
* The subject has previously been diagnosed with hepatocellular carcinoma.
* The subject has acute or exacerbating hepatitis, fluctuating or rapidly deteriorating hepatic function
* The subject has a history of drug misuse within 6 months prior to screening or a positive drug test at screening or on Day -1.
* The subject has evidence of current or recent abuse of alcohol
* The subject has received therapy known to exacerbate hepatic impairment within 4 weeks of study drug administration.
* The subject is taking antiviral therapy for treatment of active hepatitis infection at the time of screening.

Subjects with Normal Hepatic Function

* The subject has evidence of clinically significant hepatic illness or abnormalities.
* The subject has evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at screening or baseline.
* The subject tests positive for Hepatitis B virus (HBV), HBsAg, Hepatitis C virus (HCV), or Hepatitis C antibody
* The subject has used any prescription or nonprescription drugs, including over-the-counter (OTC) medications or vitamins, within 2 weeks prior to the first dose, unless otherwise specified.
* The subject has a history of drug or alcohol misuse within 6 months prior to screening or a positive drug test at screening or on Day -1.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
AUC0-t | From Day 1 to Day 7
  Area under the plasma concentration-time curve from time 0 to time of the last measurable concentration
AUC0-inf | From Day 1 to Day 7
  Area under the plasma concentration-time curve from time 0 to infinity (if data permit)
Cmax | From Day 1 to Day 7
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events as assessed by NCI CTCAE v5.0 | From Day 1 to Day 7
  To evaluate the safety of a single dose of 250mg surufatinib administered in subjects with mild (if enrolled) and moderate hepatic impairment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Orange County Research Center, Tustin, California
  - Orlando Clinical Research Center, Inc., Orlando, Florida